CLINICAL TRIAL: NCT05037513
Title: Integrated PrEP Interventions for People Who Inject Drugs in Rural Kentucky
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilary L Surratt, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Hilary L Surratt, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67933; R34DA053140 (NIH)
Record Dates: First submitted 2021-08-05; First posted 2021-09-08 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDC-PrEP (Active Comparator): 1 session PrEP education following CDC guidelines delivered one on one by an Advanced Practice Registered Nurse to individual clients in the syringe service program setting
  Interventions: Behavioral: CDC-PrEP
- SBCM-PrEP (Experimental): Multi-session Strengths-Based Case Management intervention adapted for PrEP related educational content delivered one on one by an Advanced Practice Registered Nurse to individual clients in the syringe service program setting
  Interventions: Behavioral: SBCM-PrEP

INTERVENTIONS:
Behavioral: SBCM-PrEP — Multi-session SBCM intervention adapted for PrEP initiation focus
  Arms: SBCM-PrEP
Behavioral: CDC-PrEP — 1 session PrEP education following CDC guidelines
  Arms: CDC-PrEP

SUMMARY:
The overarching goal of this study is to adapt and feasibility test an evidence-based strengths-based case management (SBCM) intervention for pre-exposure prophylaxis (PrEP) initiation, and examine preliminary efficacy of the intervention comparators (SBCM-PrEP) and (Centers for Disease Control (CDC)-PrEP). Within this context, the Specific Aims are to: 1) Assess client, provider, organization, and structural-level facilitators and barriers to integration of a PrEP focused SBCM (SBCM-PrEP) intervention into routine syringe service program (SSP) practice; 2) Adapt an evidence-based SBCM protocol to provide PrEP intervention services for people who inject drugs (PWID) in SSP sites; and, 3) Examine feasibility, acceptability and preliminary efficacy of the adapted SBCM-PrEP. 80 participants will be randomized into: CDC-PrEP (an in-use PrEP intervention based on CDC guidelines) or SBCM-PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* HIV-negative status;
* Past month drug injection;
* Client of SSP in targeted sites

Exclusion Criteria:

• HIV-positive status

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary L Surratt, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Surratt HL, Yeager HJ, Adu A, Gonzalez EA, Nelson EO, Walker T. Pre-Exposure Prophylaxis Barriers, Facilitators and Unmet Need Among Rural People Who Inject Drugs: A Qualitative Examination of Syringe Service Program Client Perspectives. Front Psychiatry. 2022 May 30;13:905314. doi: 10.3389/fpsyt.2022.905314. eCollection 2022. PMID 35706473
- [Result] Surratt HL, Brown S, Burton AL, Cranford W, Green C, Mersch SM, Rains R, Westgate PM. Examining HIV pre-exposure prophylaxis (PrEP) acceptability among rural people who inject drugs: predictors of PrEP interest among syringe service program clients. AIDS Care. 2024 Dec;36(12):1858-1868. doi: 10.1080/09540121.2024.2390067. Epub 2024 Aug 13. PMID 39137923
- [Result] Surratt HL, Brown S, Burton AL, Cranford W, Fanucchi LC, Green C, Mersch SM, Rains R, Westgate PM. Outcomes of a pilot randomized clinical trial testing brief interventions to increase HIV pre-exposure prophylaxis uptake among rural people who inject drugs attending syringe services programs. Ther Adv Infect Dis. 2025 Jan 29;12:20499361251314766. doi: 10.1177/20499361251314766. eCollection 2025 Jan-Dec. PMID 39886694

RESULTS

PARTICIPANT FLOW:
Period: Intervention Period
Arm/Group | CDC-PrEP | SBCM-PrEP
Started | 39 | 41
Completed | 38 | 39
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: Follow Up Period
Arm/Group | CDC-PrEP | SBCM-PrEP
Started | 39 | 41
Completed | 19 | 17
Not Completed | 20 | 24
Not completed — Lost to Follow-up | 16 | 21
Not completed — Death | 0 | 1
Not completed — Incarcerated | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDC-PrEP | SBCM-PrEP | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (8.6) | 39.0 (9.8) | 39.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 35 | 40 | 75
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Initiating PrEP
Description: Documented PrEP initiation, measured by dispensed PrEP prescription.
Time Frame: 3 months post-baseline
Population: We analyzed both the intent to treat (ITT) and per protocol populations. Per protocol is reported here, which includes those with any exposure to the respective interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | CDC-PrEP | SBCM-PrEP
Number analyzed (Participants) | 38 | 39
Participants | 1 | 6
Statistical Analysis 1: Comparison: CDC-PrEP vs SBCM-PrEP; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 7.06, 95% CI 2-sided [0.8 to 62.2]

2. Primary Outcome: Number of Participants Initiating PrEP
Description: Documented PrEP initiation, measured by dispensed PrEP prescription.
Time Frame: 6 months post-baseline
Population: We analyzed intent to treat (ITT) and per protocol populations. Per protocol is reported here, which includes all participants with any exposure to their respective intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | CDC-PrEP | SBCM-PrEP
Number analyzed (Participants) | 38 | 39
Participants | 1 | 6
Statistical Analysis 1: Comparison: CDC-PrEP vs SBCM-PrEP; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 7.06, 95% CI 2-sided [0.8 to 62.2]

3. Secondary Outcome: Level of Intervention Engagement Assessed by Session Checklist
Description: 5 item Session Checklist completed by Interventionist post-session; range is 5-20, lower scores are higher engagement
Time Frame: 8 weeks post-baseline
Population: Intervention engagement measure using the session checklist was collected only on the experimental arm; session checklist ratings are part of the SBCM-PrEP post session checklist forms only per study protocol, administration was planned post each of the 5 offered sessions. One SBCM-PrEP participant is missing data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDC-PrEP | SBCM-PrEP
Number analyzed (Participants) | 0 | 38
units on a scale |  | 8.68 (2.96)

4. Secondary Outcome: Level of Intervention Satisfaction Assessed by the IAQ
Description: 10 item Intervention Acceptability Questionnaire (IAQ) completed by participants post-intervention; range is 10-50, lower scores are higher acceptability
Time Frame: 8 weeks post-baseline
Population: IAQ acceptability measures were collected from the experimental SBCM-PrEP arm only as part of the post-intervention session forms per protocol. The IAQ is a descriptive measure of acceptability of the newly adapted intervention, not planned for cross-arm comparative analysis. The IAQ is a participant-completed paper survey given to participants post-session to complete independently, which accounts for the high level of missingness; many participants did not return the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDC-PrEP | SBCM-PrEP
Number analyzed (Participants) | 0 | 14
units on a scale |  | 13.2 (3.07)

ADVERSE EVENTS:
Time Frame: Participant level adverse events were collected over 6 months
Description: Adverse events were generally collected during the course of follow-up assessments using standard study instrumentation. For participants lost to follow-up, study staff collected information on deaths through publicly available information.
Arm/Group | CDC-PrEP | SBCM-PrEP
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDC-PrEP (N=39) | SBCM-PrEP (N=41)
Death (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Small sample size on the pilot was not sufficiently powered to determine efficacy, however, percent difference and effect size estimates were determined as intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT05037513/Prot_SAP_ICF_001.pdf